CLINICAL TRIAL: NCT04255368
Title: Effect of Choline Source and Gut Microbiota Composition on Trimethylamine-N-oxide Response in Humans
Brief Title: Choline Source, Gut Microbiota and Trimethylamine-N-oxide Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 8547
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Metabolism
Keywords: Dietary precursor; Metabolism; Gut microbiota

STUDY DESIGN:
Intervention Model Description: Randomized, controlled crossover design where participants consume 3 meals containing (i) free choline; (ii) phosphatidylcholine; or (iii) no choline in a random order separated by a 1-week washout period
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water-soluble choline (Experimental): A breakfast meal consisting of 1 cup of tomato soup containing 600 mg choline as choline bitartrate; served with a bagel with margarine-butter spread and one cup of water.
  Interventions: Other: Water-soluble choline
- Fat-soluble choline (Experimental): A breakfast meal consisting of 1 cup of tomato soup containing 600 mg choline as phosphatidylcholine; served with a bagel with margarine-butter spread and one cup of water.
  Interventions: Other: Fat-soluble choline
- No choline (Active Comparator): A breakfast meal consisting of 1 cup of tomato soup containing no choline; served with a bagel with margarine-butter spread and one cup of water.
  Interventions: Other: No choline control

INTERVENTIONS:
Other: Water-soluble choline — 600 mg choline as choline bitartrate
  Arms: Water-soluble choline
Other: Fat-soluble choline — 600 mg choline as phosphatidylcholine
  Arms: Fat-soluble choline
Other: No choline control — No choline
  Arms: No choline

SUMMARY:
The purpose of this research is to determine the production of trimethylamine-N-oxide (TMAO) from different forms of choline and whether this response is modified by the gut microbiota composition.

DETAILED DESCRIPTION:
The overall goal of this research is to identify dietary and physiological factors contributing to elevated levels of trimethylamine-N-oxide (TMAO), a choline-derived gut-microbiome-dependent metabolite that has been identified to increase cardiovascular disease risk. Our recent findings indicate that the gut microbiome may account for variations in TMAO levels, whereby those with a greater enrichment of Firmicutes to Bacteroidetes had elevated TMAO response to dietary precursor intake. However, the interaction between choline intake and gut microbiota composition as a determinant of interindividual variations in TMAO response has not been investigated. This study sought to i) compare plasma and urinary TMAO response after acute challenge containing different forms of choline; and ii) to determine the association between differences in TMAO response with differences in gut microbiota composition. To accomplish these objectives, a randomized, controlled cross-over study was conducted in healthy participants (n=41). The study incorporated three arms comprised of study meals containing (i) 600 mg choline as choline bitartrate; (ii) 600 mg choline as phosphatidylcholine; or (iii) no choline. Each meal was served with a bagel with margarine-butter spread and one cup of water, administered in a single day and separated by a 1-week washout period. Baseline blood sample was obtained by a phlebotomist using a standard venipuncture procedure, and participants collected their baseline urine sample. They also turned in a one-time self-collected baseline stool sample. Following the consumption of the study meal, serial blood samples were collected at 30 min and 1, 2, 4 and 6 h, and urine samples collected throughout the 6 h study period. At 4.5 h, participants were provided a fixed fruit snack (i.e., 2 single serving prepackaged applesauce) and water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of any race or ethnicity
* Age 21-50 y
* BMI 20-24.9 kg/m2 or BMI 30-39.9 kg/m2

Exclusion Criteria:

* Age > 50 y
* BMI outside of the normal-weight or obese range (BMI < 20 kg/m2; BMI 25-29.9 kg/m2; or BMI > or = 40 kg/m2)
* Pregnant or planning to become pregnant during the course of the study; currently breastfeeding (females)
* Vegetarians
* Smokers or recreational drug users
* Individuals with gastrointestinal diseases or complaints, chronic illnesses or other metabolic diseases (including trimethylaminuria)
* Individuals who have taken antibiotics within the past 2 months
* Individuals who are not willing to discontinue pre- and probiotics and dietary supplements for the time leading up to 2 months before the study and during the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
TMAO metabolite concentration change | Blood: study baseline, 30 minutes and 1 hour, 2 hours, 4 hours and 6 hours
  Plasma TMAO metabolite response
TMAO metabolite concentration change | Urine: study baseline, pooled 6 hours study period
  Urinary TMAO metabolite response
Gut microbiome profile | Stool: one-time baseline
  16S rRNA

SECONDARY OUTCOMES:
One-carbon metabolite concentration change | Blood: study baseline, 30 minutes and 1 hour, 2 hours, 4 hours and 6 hours
  Plasma choline metabolite response
Phosphatidylcholine concentration change | Blood: study baseline, 30 minutes and 1 hour, 2 hours, 4 hours and 6 hours
  Plasma phosphatidylcholine response
One-carbon metabolite concentration change | Urine: study baseline, pooled 6 hours study period
  Urinary choline metabolite response
Inflammation and cardiovascular disease risk marker concentration change | Blood: study baseline to 6 hours
  Plasma TNF-α and IL-6
Flavin monooxygenase 3 (FMO3) 472 G>A genotype variant | Blood: study baseline
  Genetic polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Clara E Cho, PhD, Principal Investigator — Utah State University
Locations (1):
- Center for Human Nutrition Studies Clinic, Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Cho CE, Taesuwan S, Malysheva OV, Bender E, Tulchinsky NF, Yan J, Sutter JL, Caudill MA. Trimethylamine-N-oxide (TMAO) response to animal source foods varies among healthy young men and is influenced by their gut microbiota composition: A randomized controlled trial. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600324. Epub 2016 Aug 3. PMID 27377678